CLINICAL TRIAL: NCT02466633
Title: Effect of Monitoring System Design on Response Time to Cardiac Arrhythmias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00053941; 1R01HS023387-01 (AHRQ)
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Change in in-hospital cardiac monitoring method (Experimental): Pre- and post-intervention, where the intervention is a change in in-hospital cardiac monitoring method
  Interventions: Other: In-hospital cardiac monitoring method

INTERVENTIONS:
Other: In-hospital cardiac monitoring method — Method for monitoring hospitalized patients at risk for cardiac arrhythmias (non-ICU)

SUMMARY:
To increase the potential for timely detection and treatment of cardiac events, hospitals have implemented a number of different cardio-respiratory monitoring methods for at-risk patients. The goal of this study is to compare different monitoring methods to determine the most efficient method to monitor hospitalized patients - the method that will lead to the quickest response to critical heart rhythms. The investigators will then test the efficiency of this monitoring method by implementing it in a new patient care unit.

DETAILED DESCRIPTION:
Most patients in the hospital who are at lower risk for developing abnormal heart rhythms have their vitals signs (e.g., heart rate, blood pressure) measured intermittently, such as every 8 hours. In contrast, hospitalized patients who are at risk for cardiac arrest and other arrhythmias are put on telemetry to continuously monitor their heart rhythm. A telemetry monitor is a portable box that is attached to the patient's ECG leads and displays his or her heart rate and rhythm at a central station. The monitor sends an alarm when it detects an abnormal rhythm, notifying the person monitoring the patient to check on the patient. Monitor watchers are dedicated nurses or technicians who monitor a bank of displays . The watcher-to-patient ratio varies among hospitals, with a single watcher monitoring between 16 and 72 patients at one time. There are also variations in the additional tasks assigned to watchers, communication modalities between watchers and nurses (e.g., pagers, overhead speakers, landline and cell phones, or bi-directional voice communication badges), and alarm presentation to nurses (e.g., via bedside monitors, centrally located monitors, automated phone notifications, or none at all, relying on telemetry watchers for notifications).

A quick and efficient response to cardiac arrest is critical in order to increase the patient's chance of survival. There is a need for a better understanding of the impact on monitoring efficiency of factors such as the workload of monitor watchers, communication methods, and supportive technologies including alarms and automated notification systems. The objective of the proposed research is to identify and test determinants of efficient cardiac monitoring methods. There are 3 phases to the study:

1. Characterize candidate monitoring methods (Phase 1). The investigators will study usual care for monitored patients in 6 hospital units. As part of their usual care these units have different monitoring methods. These methods vary in terms of 1) the location of the monitor watchers, 2) the means of communicating routine and life-threatening events (e.g., via pagers), and 3) monitor watchers' patient load and workload. For each of these 6 units, the investigators will collect data through interviews, observations, and 20 cardiac arrest simulations.
2. Determine which monitoring method leads to consistently rapid response times to lethal arrhythmias (Phase 2). Using interview, observation, and simulation data collected in Phase 1, the investigators will develop a computer simulation model of each of the 6 monitoring methods that will allow them to identify the most efficient method.
3. Test a new monitoring method (Phase 3). In one of the units we had previously conducted arrhythmia simulations, we will conduct 20 additional simulations after a change from remote telemetry monitoring to local nurse-based monitoring. We will evaluate whether response times decrease with the new monitoring method.

ELIGIBILITY:
Inclusion Criteria:

* Care providers including the individuals responsible for monitoring patients (monitoring technicians and nurses), individuals communicating life threatening events (monitoring technicians, health unit coordinators, and nurses) and the individuals responsible for the initial check on a patient in the event of life-threatening cardiac arrhythmias (generally the patient's nurse).
* Patients for whom cardiac monitoring was ordered by their physician.

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Response time to a simulated (not real) critical cardiac arrhythmia (pulseless ventricular tachycardia or ventricular fibrillation) | After critical arrhythmia is simulated (approximately 1-5 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Noa Segall, PhD, Principal Investigator — Duke University